CLINICAL TRIAL: NCT06140290
Title: A PHASE 1, OPEN-LABEL, SINGLE DOSE, FIXED-SEQUENCE CROSSOVER SUB STUDY TO DETERMINE THE PHARMACOKINETICS USING TASSO DEVICE AND SAFETY AND TOLERABILITY USING WEARABLE MONITORING DEVICES FOLLOWING SINGLE ORAL DOSES OF ETRASIMOD 2 MG IR TABLETS IN HEALTHY ADULT PARTICIPANTS IN A HYBRID DECENTRALIZED CLINICAL TRIAL DESIGN
Brief Title: A Sub Study to Evaluate the Study Medication (Etrasimod) Using Wearable Sensors in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5041050; C5041034 Sub-Study (Other: Alias Study Number); 2023-508119-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: etrasimod; adults
MeSH Terms: interventions — etrasimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fixed Sequence (Experimental): Single oral dose of etrasimod 2mg tablet under fasted conditions with site staff led assessments and training on how to use wearable sensors followed by single oral dose 2mg tablet under fasted conditions with participant led assessments with wearable sensors.
  Interventions: Drug: Etrasimod Immediate Release (IR)

INTERVENTIONS:
Drug: Etrasimod Immediate Release (IR) — An immediate release tablet

SUMMARY:
The purpose of this study is to look at how healthy adults process Etrasimod when assessed by wearable sensors. Etrasimod is taken without food and assessments taken by site staff and then by participants after training.

The study is seeking participants who are:

* Aged 18 or older
* Male or female who are healthy as determined by medical assessment
* Body-mass index (BMI) of 16 to 32, and a total body weight > 50kg.

The study will take up to 9 weeks, including the screening period. Participants will have to stay at the study clinic for at least 2 nights, in each of 2 study periods.

Participants will take Etrasimod as a tablet by mouth without food. Blood samples will be taken both before and after participants take Etrasimod. Participants will also use wearable devices to assess blood pressure, heart rate and take further blood samples. A follow-up phone call will be made 20 to 27 days after the last study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* BMI 16 to 32 kg/m2
* body weight more than 50kg

Exclusion Criteria:

* Ongoing or past history of significant medical conditions
* Eye disorders such as macular edema or uveitis
* Ongoing or recent infections
* Use of prescription or non prescription medications within 7 days of first dose
* Smoking or using nicotine products equivalent to more than 5 cigarettes per day
* History of severe allergic or anaphylactic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants were enrolled in this present study.
Pre-assignment Details: For secondary pharmacokinetic (PK) outcome measures' analysis, as planned, data of participants who received Etrasimod 2 mg IR tablet (Treatment A) in C5041034 study [NCT05956002] is used for comparison. These participants were not enrolled in the present study C5041050 [NCT06140290], only the relevant historical data was used for comparison as per the objectives.
Groups:
- Period 1: Etrasimod 2mg (Treatment F, With Practice Session): Participants received a single oral dose of Etrasimod 2 milligram (mg) immediate release (IR) with 240 milliliter (mL) water under fasting conditions on Day 1 of Period 1 (Treatment F). Participant were given practice sessions on Tasso and wearable monitoring devices on Day 2.
- Period 2: Etrasimod 2mg (Treatment G, Without Practice Session): Participants received a single oral dose of Etrasimod 2 mg IR tablet with 240 mL water under fasting conditions on Day 1 of Period 2 (Treatment G). Participants were not given practice sessions on Tasso and wearable monitoring devices.
Period: Period 1
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Started | 8 | 0
Treated | 8 | 0
Completed | 7 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Started | 0 | 8
Treated | 0 (Period 2 was followed by Period 1. Participants entered from Period 1 to Period 2.) | 7 (Period 2 was followed by Period 1. Participants entered from Period 1 to Period 2.)
Completed | 0 | 6
Not Completed | 0 | 2
Not completed — Assigned but not treated | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who took at least 1 dose of study intervention.
Groups:
- All Participants: Etrasimod 2mg: All participants who received study treatment either in Period 1 or 2 of the study.
Arm/Group | All Participants: Etrasimod 2mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-Time Profile From Time Zero to 24 Hours (AUC0-24) of Etrasimod: Tasso PK Sampling
Description: AUC0-24 was calculated as linear/log trapezoidal method. PK sampling: a) Treatment F/Reference: Tasso PK micro sampling was done by clinical research unit (CRU) staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 1 of each period
Population: PK parameter analysis set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL )
Groups:
- Period 1: Etrasimod 2mg (Treatment F, With Practice Session): Participants received a single oral dose of Etrasimod 2 mg IR with 240 mL water under fasting conditions on Day 1 of Period 1 (Treatment F). Participant were given practice sessions on Tasso and wearable monitoring devices on Day 2.
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Nanogram*hour per milliliter (ng*hr/mL ) | 666.4 (23) | 745.5 (25)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Period 2: Etrasimod 2mg (Treatment G, Without Practice Session); Analysis was performed using a mixed effect model, with treatment as a fixed effect and participant as a random effect; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Here, Etrasimod 2mg (Treatment F) with practice session was the reference treatment, while Etrasimod 2mg (Treatment G) without practice session was the test treatment; Ratio of Adjusted Geometric Means = 108.32, 90% CI 2-sided [101.20 to 115.94] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

2. Primary Outcome: Area Under the Serum Concentration-Time Profile From Time 24 Hours to the Time of the Last Quantifiable Concentration (AUC24hr-last) of Etrasimod: Tasso PK Sampling
Description: AUC24hr-last was calculated as linear/log trapezoidal method. PK sampling: a) Treatment F/Reference: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely.
Time Frame: 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: PK parameter analysis set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 6
ng*hr/mL | 768.4 (37) | 872.1 (16)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Period 2: Etrasimod 2mg (Treatment G, Without Practice Session); Analysis was performed using a mixed effect model, with treatment as a fixed effect and participant as a random effect; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 120.41, 90% CI 2-sided [108.02 to 134.22] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

3. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Etrasimod: Tasso PK Sampling
Description: AUCinf was calculated as AUClast + (Clast*/kel), where AUClast is area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast). Clast is the predicted plasma concentration at the last quantifiable time point and Kel is the terminal phase rate constant. PK sampling: a) Treatment F/Reference: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 6
ng*hr/mL | 1503 (32) | 1652 (19)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Period 2: Etrasimod 2mg (Treatment G, Without Practice Session); Analysis was performed using a mixed effect model, with treatment as a fixed effect and participant as a random effect; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 115.29, 90% CI 2-sided [105.17 to 126.38] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

4. Primary Outcome: Maximum Observed Concentration (Cmax) of Etrasimod: Tasso PK Sampling
Description: PK sampling: a) Treatment F/Reference: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Nanogram per milliliter (ng/mL) | 40.65 (26) | 44.63 (28)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Period 2: Etrasimod 2mg (Treatment G, Without Practice Session); Analysis was performed using a mixed effect model, with treatment as a fixed effect and participant as a random effect; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Adjusted Geometric Means = 106.75, 90% CI 2-sided [99.33 to 114.73] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

5. Secondary Outcome: AUC0-24 of Etrasimod: Tasso and Venous PK Sampling
Description: AUC0-24 was calculated as linear/log trapezoidal method. In this outcome measure, as planned, data of participants who received Etrasimod 2 mg IR tablet (Treatment A) in C5041034 study is used for comparison. PK sampling: a) Treatment F/Test: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely; c) Treatment A/Reference: Venous PK sampling from pre-dose (0 hour) till 168 hours post-dose.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study: Participants who received a single oral dose of Etrasimod 2 mg IR tablet with 240 mL of water on Day 1 of Period 1, 2, 3 or 4 under fasting conditions (Treatment A) in the study C5041034. Only the relevant historical data from these participants is utilized, they are not enrolled in the present study.
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) | Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study
Number analyzed (Participants) | 8 | 7 | 16
ng*hr/mL | 666.4 (23) | 745.5 (25) | 725.8 (21)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA (Analysis of variance) model with treatment as a fixed effect; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Here, Etrasimod 2mg (Treatment F) with practice session was the test treatment, while Etrasimod 2mg IR tablet (Treatment A) was the reference treatment; Ratio of Adjusted Geometric Means = 91.80, 90% CI 2-sided [77.76 to 108.38] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages
Statistical Analysis 2: Comparison: Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Here, Etrasimod 2mg (Treatment G) without practice session was the test treatment, while Etrasimod 2mg IR tablet (Treatment A) was the reference treatment; Ratio of Adjusted Geometric Means = 102.71, 90% CI 2-sided [86.33 to 122.19] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

6. Secondary Outcome: AUC24hr-last of Etrasimod: Tasso and Venous PK Sampling
Description: AUC24hr-last was calculated as linear/log trapezoidal method. In this outcome measure, as planned, data of participants who received Etrasimod 2 mg IR tablet (Treatment A) in C5041034 study is used for comparison. PK sampling: a) Treatment F/Test: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely; c) Treatment A/Reference: Venous PK sampling from pre-dose (0 hour) till 168 hours post-dose.
Time Frame: 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) | Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study
Number analyzed (Participants) | 8 | 6 | 16
ng*hr/mL | 768.4 (37) | 872.1 (16) | 890.1 (31)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Ratio of Adjusted Geometric Means = 86.34, 90% CI 2-sided [69.42 to 107.37] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages
Statistical Analysis 2: Comparison: Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Ratio of Adjusted Geometric Means = 97.98, 90% CI 2-sided [76.99 to 124.70] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

7. Secondary Outcome: AUCinf for Etrasimod: Tasso and Venous PK Sampling
Description: AUCinf was calculated as AUClast + (Clast*/kel), where AUClast is area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast). Clast is the predicted plasma concentration at the last quantifiable time point and Kel is the terminal phase rate constant. PK sampling: a) Treatment F/Test: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely. c) Treatment A/Reference: Venous PK sampling from pre-dose (0 hour) till 168 hours post-dose.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) | Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study
Number analyzed (Participants) | 8 | 6 | 16
ng*hr/mL | 1503 (32) | 1652 (19) | 1694 (26)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Ratio of Adjusted Geometric Means = 88.72, 90% CI 2-sided [73.10 to 107.68] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages
Statistical Analysis 2: Comparison: Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Ratio of Adjusted Geometric Means = 97.54, 90% CI 2-sided [78.74 to 120.83] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

8. Secondary Outcome: Cmax for Etrasimod: Tasso and Venous PK Sampling
Description: PK sampling: a) Treatment F/Test: Tasso PK micro sampling was done by CRU staff participants at the CRU up to 24 hours post-dose and by participants 48-168 hours post-dose remotely; b) Treatment G/Test: Tasso PK micro sampling was done by participants at the CRU up to 24 hours post-dose and 48-168 hours post-dose remotely. c) Treatment A/Reference: Venous PK sampling from pre-dose (0 hour) till 168 hours post-dose.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) | Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study
Number analyzed (Participants) | 8 | 7 | 16
ng/mL | 40.65 (26) | 44.63 (28) | 43.18 (22)
Statistical Analysis 1: Comparison: Period 1: Etrasimod 2mg (Treatment F, With Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Ratio of Adjusted Geometric Means = 94.14, 90% CI 2-sided [79.01 to 112.17] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages
Statistical Analysis 2: Comparison: Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) vs Etrasimod 2mg IR Tablet: Treatment A, C5041034 Study; Analysis was performed using ANOVA model with treatment as a fixed effect; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Ratio of Adjusted Geometric Means = 103.36, 90% CI 2-sided [86.04 to 124.16] — Ratio (Test/Reference) and its associated 90% CI were expressed as percentages

9. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 1, 2, 3, 4 ,5, 6, 8 and 24 Hours Post-dose on Day 1
Description: Heart rate was measured in beats per minute (beats/min). Baseline was defined as the average of triplicate electrocardiogram (ECG) HR measurements collected at pre-dose (0 hour) on Day 1 of each period.
Time Frame: Baseline; 1, 2, 3 ,4, 5, 6, 8 and 24 hours post-dose on Day 1 of each period
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Beats/minute
  Change at 1 hour | -4.9 (3.56) | -3.4 (1.72)
  Change at 2 hours | -10.8 (4.33) | -10.3 (2.75)
  Change at 3 hours | -10.8 (5.44) | -10.9 (2.34)
  Change at 4 hours | -10.8 (5.73) | -10.1 (3.44)
  Change at 5 hours | -4.6 (4.44) | -2.4 (3.46)
  Change at 6 hours | -7.0 (5.58) | -2.0 (5.92)
  Change at 8 hours | -9.0 (6.82) | -4.9 (4.56)
  Change at 24 hours | -8.4 (4.60) | -1.9 (5.01)

10. Secondary Outcome: Change From Baseline to Nadir in HR at Day 1
Description: Heart rate was measured in beats per minute (beats/min). Baseline was defined as the average of triplicate ECG HR measurements collected at pre-dose (0 hour) on Day 1 of each period. Nadir HR was taken as the minimum HR from all ECGs taken post-Etrasimod on day 1 of each period. If Nadir HR was attained at multiple post-dose time points on Day 1, only the latest time point was summarized.
Time Frame: Baseline; Anytime or latest time with minimum HR measurement taken post-dose on Day 1 of each period
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Beats/ min
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Beats/ min | -14.1 (5.14) | -12.1 (2.27)

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred on or after the first dose of study treatment up to 35 days post last dose of study treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect.
Time Frame: Day 1 up to 35 days after last dose of study treatment (maximum up to 45 days)
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Participants | 7 | 5

12. Secondary Outcome: Number of Participants With Clinically Significant Findings in Laboratory Abnormalities
Description: Clinical laboratory abnormalities test criteria included, a) hematology: lymphocytes (10^3/millimeter [mm)^3]) and lymphocytes/leukocytes percentage (%) less than (<) 0.8* lower limit of normal (LLN), eosinophils (10^3/mm^3), eosinophils/leukocytes (%) and monocytes (10^3/mm^3) greater than (>)1.2* upper limit of normal (ULN); b) Urinalysis: urine glucose, ketones, urine hemoglobin and bilirubin, leukocyte esterase greater than equal to (>=) 1. Clinical significance of laboratory abnormalities was determined by the investigator.
Time Frame: Day 1 up to 35 days after last dose of study treatment (maximum up to 45 days)
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Vital signs included blood pressure systolic and diastolic millimeter of mercury (mmHg) and pulse rate (beats/min). Clinical significance of vital signs abnormalities was determined by the investigator.
Time Frame: Day 1 up to 35 days after last dose of study treatment (maximum up to 45 days)
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination
Description: A complete physical examination test included, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief physical examination test included, at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant reported symptoms. Clinical significance of physical examination abnormalities was determined by the investigator.
Time Frame: Day 1 up to 35 days after last dose of study treatment (maximum up to 45 days)
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Participants | 0 | 0

15. Secondary Outcome: Number of Participants Categorized Per Pre-defined Electrocardiogram (ECG) Findings Criteria
Description: ECG findings criteria for QT interval corrected using Fridericia's formula (QTcF) were as: 450 millisecond (msec) < value less than equal (<=) 480 msec, 480 msec < value <=500 msec, >500 msec, 30 msec <= change from baseline <=60 msec, change from baseline >60 msec.
Time Frame: From Baseline (Day 1) maximum up to Day 17
Population: SAS included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
Number analyzed (Participants) | 8 | 7
Participants
  450 msec < Value <= 480 msec | 1 | 0
  480 msec < Value <= 500 msec | 0 | 0
  Value > 500 msec | 0 | 0
  30 msec <= Change from baseline <= 60 msec | 0 | 0
  Change from baseline > 60 msec | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 35 days after last dose of study treatment (maximum up to 45 days)
Description: SAS included all participants who took at least 1 dose of study intervention.
Arm/Group | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 7/8 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Etrasimod 2mg (Treatment F, With Practice Session) (N=8) | Period 2: Etrasimod 2mg (Treatment G, Without Practice Session) (N=7)
Atrioventricular block first degree (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Application site irritation (General disorders) | 4 | 0
Influenza like illness (General disorders) | 1 | 0
Puncture site injury (General disorders) | 2 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Device issue (Product Issues) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT06140290/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT06140290/SAP_001.pdf